CLINICAL TRIAL: NCT00784745
Title: Is Insulin Resistance and/or Glucose Intolerance Pathogenetic in the Development of a Reduced Incretin Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Kasper Aaboe, Doctor, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H-D-2008-087
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Insulin Resistance; Glucose Intolerance
Keywords: incretin effect; type 2 diabetes; GLP-1; GIP; dexamethasone
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 2mg morning and night for 5 days.

SUMMARY:
The purpose of this study is to examine whether there is a causal relationship between insulin resistance and/or glucose intolerance in the development of a defect incretin effect.

DETAILED DESCRIPTION:
In this study we are going to examine the incretin effect before and after the development of insulin resistance and/or glucose intolerance. The incretin effect is the increased insulin response seen after an oral as apposed to an intravenous glucose challenge with identical plasma glucose profiles. This insulin enhancing effect is greatly reduced in type 2 diabetes.

Since the development of type 2 diabetes is preceded by insulin resistance and glucose intolerance we wanted to examine the incretin effect in the early stages of type 2 diabetes.

To do this, we want to induce insulin resistance and/or glucose intolerance. This is achieved by 5 days of treatment with dexamethasone.

The incretin effect in this study will be examined by 3 investigations prior to the treatment and 3 days following the treatment.

Day 1: Oral glucose challenge with 75 g of glucose.

The subject is asked to drink 75g of glucose suspended in 300mL of water. During the 4 hours of the test, we draw blood at various times during the study to determine the concentration of: Glucose, GLP-1, GIP, Glucagon, Insulin and c-peptide.

Day 2: Intravenous glucose

We duplicate the glucose curve obtained from day 1. We also draw blood during this test to the same end as in day 1.

Day 3: Mixed meal.

The subjects are served a mixed meal. During this 4 hour test, we draw blood to examine the response to a standardized meal. The test involves sampling blood as described for the other days.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians >20 years
* Normal glucose tolerance as assessed by the WHO criteria
* First degree relative and at least 1 second degree relative with type 2 diabetes
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT/ASAT > 2 times normal value)
* Kidney disease (S-creatinin > 130uM and/or albuminuria)
* Heart disease (NYHA II, III or IV)
* Treatment with medicine that cannot be paused
* Pregnancy of breast feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incremental GLP-1 response during the mixed meal test. Assessed as AUC during the 4 hour test. | 4 hours (during the mixed meal test)

CONTACTS AND LOCATIONS:
Overall Officials: Thure Krarup, dr. med., Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Henriksen JE, Alford F, Ward GM, Beck-Nielsen H. Risk and mechanism of dexamethasone-induced deterioration of glucose tolerance in non-diabetic first-degree relatives of NIDDM patients. Diabetologia. 1997 Dec;40(12):1439-48. doi: 10.1007/s001250050847. PMID 9447952
- [Derived] Jensen DH, Aaboe K, Henriksen JE, Volund A, Holst JJ, Madsbad S, Krarup T. Steroid-induced insulin resistance and impaired glucose tolerance are both associated with a progressive decline of incretin effect in first-degree relatives of patients with type 2 diabetes. Diabetologia. 2012 May;55(5):1406-16. doi: 10.1007/s00125-012-2459-7. PMID 22286551